CLINICAL TRIAL: NCT03056560
Title: TakeCARE: A Video Bystander Program to Prevent Sexual Violence on College Campuses
Brief Title: Evaluating a Video Bystander Program for First-Year College Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Ernest Jouriles, Professor, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R21HD085063 (NIH)
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Bystander Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Bystander Program (Experimental): TakeCARE video
  Interventions: Behavioral: TakeCARE (video bystander program)
- Control Video (No Intervention): Study Skills Video

INTERVENTIONS:
Behavioral: TakeCARE (video bystander program) — brief video encouraging active responses to high-risk situations for campus violence
  Arms: Video Bystander Program

SUMMARY:
This study will evaluate an innovative video bystander program, which has the potential to be implemented broadly and cost-effectively across college campuses. Half of the participants will receive the video bystander program, and the other half will not.

DETAILED DESCRIPTION:
Sexual violence, which includes both sexual coercion and assault, is a significant problem on college campuses due to its high prevalence and adverse consequences. This research will evaluate an innovative video bystander program, which has the potential to be implemented broadly and cost-effectively across college campuses. We will recruit first-year college students from each of 4 college campuses (Southern Methodist University, Marquette University, William Paterson University, and Stony Brook University).

The video bystander program (TakeCARE) starts with a narrator acknowledging the various demands placed on students in attempting to balance adult responsibilities with the social opportunities of college, as well as the importance of keeping safe while engaging in these social activities. The program describes how likely it is that people they know may become a victim of sexual violence and how they can help "take care of their friends" to help prevent victimization. TakeCARE includes 3 video vignettes that demonstrate ways that students can intervene when they see sexual coercion, relationship violence, or other situations that might result in harm.

After a baseline assessment, students will be randomly assigned to view one of two video programs: TakeCARE (the video bystander program) or a control video program. A post-treatment assessment will be completed within a week of viewing the video program, and follow-up assessments will be completed 2 months and 6 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* first-year college students

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Change in bystander behavior | Baseline and 2 months
  Self-report measure: Bystander Behavior Scale

SECONDARY OUTCOMES:
Change in bystander behavior | Baseline and 2 months
  Observations using virtual reality protocol
Change in bystander efficacy | Baseline and 2 months
  Self-report measure: Bystander Efficacy Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Jouriles, Ph.D., Principal Investigator — Southern Methodist University
Locations (1):
- Southern Methodist University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No